CLINICAL TRIAL: NCT01690702
Title: Neo-/Adjuvant Phase III Trial to Compare Intense Dose-dense Chemotherapy to Tailored Dose-dense Chemotherapy in Patients With High-risk Early Breast Cancer (GAIN-2)
Brief Title: Study of Nab-Paclitaxel in High Risk Early Breast Cancer
Acronym: GAIN-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Celgene (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 68
Record Dates: First submitted 2012-08-29; First posted 2012-09-24 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; tailored; high-risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; 130-nm albumin-bound paclitaxel; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dtEC-dtD (Active Comparator): Epirubicin and Cyclophosphamide with a tailored dose 4 cycles q2w followed by one additional week followed by Docetaxel with a tailored dose 4 cycles q2w.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- EnPC (Experimental): Epirubicin 150mg/qm 3 cycles q2w followed by nabPaclitaxel 260-330mg/qm (to be determined in run-in-phase) 3 cycles q2w followed by Cyclophosphamide 2000mg/qm 3 cycles q2w
  Interventions: Drug: Epirubicin; Drug: nab-Paclitaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Epirubicin
Drug: nab-Paclitaxel
  Arms: EnPC
Drug: Cyclophosphamide
Drug: Docetaxel
  Arms: dtEC-dtD

SUMMARY:
two-armed trial to compare E-nP-C against tailored dtEC-dtD in patients with high risk early breast cancer

DETAILED DESCRIPTION:
The Norton-Simon-Hypothesis on log cell kill suggests that chemotherapy should be given at maximum dosages at minimum intervals. Combination chemotherapy, which always has to make compromises regarding the doses of each drug and treatment intervals due to acute as well as cumulative toxicities, does therefore not comply with this theory. Sequential application of monotherapies, however, allows very high single agent doses and dose-dense treatment intervals. Regimens designed according to the Norton-Simon-Hypothesis have shown to be highly active as adjuvant treatment for early breast cancer. As the number of cycles of each agent can be restricted to 3, as previously done in the AGO ETC trial by Möbus et al., cumulative toxicities do not really occur.

Two large scale trials of dose-dense chemotherapy have proven very high protective activity against tumor recurrence (AGO ETC (Ref.1) and CALGB 9741 (Ref.2)). Especially the ETC trial (epirubicin, solvent-based paclitaxel, and cyclophosphamide) showed an impressive superior DFS and OS in 1284 high-risk breast cancer patients with > 4positive lymph nodes. The doses used are exceptional at maximum dosage and minimum intervals with epirubicin 150 mg/m², Paclitaxel 225 mg/m² and cyclophosphamide 2.5 g/m² given every 2 weeks based on the above described Norton-Simon-Hypothesis. However, as each drug was given only 3 times at intervals of 2 weeks, this regimen is feasible and safe with primary support of G-CSF and ESF. The ETC schedule is today considered standard of care for high-risk breast cancer patients in Germany.

However, both trials, ETC and CALGB 9741, compared the dose-dense concept against EC-P q3w which is nowadays considered to be an inferior regimen compared to EC-P weekly or EC-Doc. The GAIN trial had a 2x2 factorial design and explored ETC versus EC-TX and ibandronate vs. observation. The trial closed recruitment after 3023 pts in July 2008. In the Panther trial, a joint effort of SBG, ABCSG, AGO-B and GBG, the tailored, dose-dense EC-Doc (dtEC-dtD) regimen was tested against conventional dosed FEC-Doc. Efficacy results are to be awaited, safety results will be published in 2012.

Nab-paclitaxel (nP) provides a better toxicity profile and a higher efficacy compared to solvent based taxanes (paclitaxel and docetaxel). It might therefore be the preferred component in an intense dose-dense regimen. Assuming that the corresponding dose of nab-paclitaxel to 175 mg/m² paclitaxel is 260 mg/m², an appropriate dose would be 330 mg/m² nab-paclitaxel to substitute paclitaxel at 225 mg/m². So far, no experience with such a dose of nab-paclitaxel is available. However, initial experience with 300mg/m² q3w and 150mg/m² weekly (in 3 out of 4 weeks) showed a good safety profile even when given for a median of 8 cycles (Ref.3). Another pilot study showed a good tolerability of 260 mg/m² nab-paclitaxel given q2w for 4 cycles (Ref.4+5).

The GAIN-2 trial will allow for comparing the toxicity and effectiveness of a predefined intense dose-dense regimen (EnPC) vs. a dose-dense regimen with modification of single doses depending on individual haematological and non-haematological toxicities. The primary aim of the GAIN-2 trial will be to compare the invasive disease-free survival after adjuvant chemotherapy with EnPC or dtEC-dtD in patients with primary node-positive or high risk node negative breast cancer. To explore the maximum dose of nab-paclitaxel in this setting, a run-in phase with varying doses of nab-paclitaxel is included in the study design.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Histologically confirmed unilateral or bilateral primary carcinoma of the breast.
3. Age at diagnosis at least 18 years, female, and biologically not older than 65 years (but in any case not older than 70 years).
4. In case of adjuvant therapy: Adequate surgical treatment with histological complete resection (R0) of the invasive breast tumor. Choice of axilla surgery is up to the participating site.
5. Centrally confirmed ER/PgR/HER2 and Ki-67 status detected on surgical removed tissue (for adjuvant patients) or from core biopsy (for neoadjuvant patients). ER/PR positive is defined as ≥ 1% stained cells and HER2 positive is defined as IHC 3+ in > 10% immunoreactive cells or FISH (or equivalent test) ratio ≥ 2.0. Formalin-fixed, paraffin-embedded (FFPE) breast tissue has to be sent to the Institute of Pathology at the Charité Berlin prior to randomization.
6. High risk breast cancer as defined as:

   * HER2 positive or triple-negative tumors irrespective of nodal status or
   * Luminal B-like tumors (ER and/or PgR positive, HER2 negative, Ki-67 > 20%) with involved lymph nodes or
   * 4 or more involved lymph nodes.
7. Complete staging work-up within 3 months prior to randomization. All patients must have performed bilateral mammography, breast ultrasound, breast MRT (optional), chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRT and bone scan. In case of positive bone scan, bone X-ray (or CT or MRT) is mandatory. Other tests may be performed as clinically indicated.
8. Karnofsky Performance status index ≥ 80%.
9. Estimated life expectancy of at least 10 years irrespective of the diagnosis of breast cancer.
10. Confirmed normal cardiac function by ECG and cardiac ultrasound (LVEF or shortening fraction) within 2 weeks prior to randomization. LVEF must be above 55%.
11. Laboratory requirements:

    Hematology
    * Absolute neutrophil count (ANC) ≥ 2.0 x 109/L and
    * Platelets ≥ 100 x 109/L and
    * Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L). Hepatic function
    * Total bilirubin ≤ 1.5x above upper normal limits (UNL) and
    * ASAT (SGOT) and ALAT (SGPT) ≤ 1.5x UNL and
    * Alkaline phosphatase ≤ 2.5x UNL. Renal function Creatinine ≤ 1.25 UNL,
    * Creatinine Clearance > 30mL/min (if creatinine is above UNL, according to Cockroft-Gault).
12. Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential.
13. Complete baseline documentation must be submitted via MedCODES and approved by GBG Forschungs GmbH.
14. Patients must be available and compliant for central diagnostics, treatment and follow-up.

Exclusion Criteria:

1. Patients with Luminal A-like tumors (ER and or PgR positive, HER2 negative and Ki-67 ≤ 20%) and

   * if neoadjuvant: < cN2 or < pN2(sn).
   * if adjuvant: < 4 involved lymph nodes.
2. Non-operable breast cancer.
3. In case of adjuvant therapy: time since axillary dissection or SLNB > 3 months (optimal < 1 month).
4. Previous and already (neoadjuvant or adjuvant) treated invasive breast carcinoma.
5. Previous malignant disease being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
6. Known or suspected congestive heart failure (> NYHA I) and/or coronary heart disease, angina pectoris requiring anti-anginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP > 160/90mm Hg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
7. Evidence for infection including wound infections, HIV, hepatitis.
8. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
9. Pre-existing motor or sensory neuropathy of a severity ≥ grade 1 by NCI-CTCAE version 4.0.
10. Other severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study.
11. Previous or concurrent treatment with:

    * concurrent chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (≤ 10mg methylprednisolone or equivalent) except inhalative corticoids.
    * concurrent sex hormones. Prior treatment must be stopped before study entry.
    * concurrent treatment with any investigational, not marketed drug within 30 days prior to study entry.
    * previous or concurrent anti-cancer therapy for any reason.
12. Absolute contraindications for the use of corticosteroids.
13. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.
14. Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2886 (Actual)
Dates: Start 2012-09; Primary Completion 2018-09-30 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
invasive disease-free survival (IDFS) | 5 years
  The IDFS is defined as the time period between the registration and the first invasive event. It will be analyzed after the end of the study by referring to data from GBG patient's registry.

SECONDARY OUTCOMES:
locoregional relapse-free survival (LRRFS) | 5 years
  The LRRFS is defined as the time period between the registration and the first locoregional event. It will be analyzed after the end of the study by referring to data from GBG patient's registry.
overall survival (OS) | 5 years
  The OS is defined as the time period between the registration and the death of a patient. It will be analyzed after the end of the study by referring to data from GBG patient's registry (relatives can give the information regarding death as well).
distant disease-free survival (DDFS) | 5 years
  The DDFS is defined as the time period between the registration and the first distant event. It will be analyzed after the end of the study by referring to data from GBG patient's registry.
local relapse-free survival (LRFS) | 5 years
  LRFS is defined as the time period between registration and first local event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
regional relapse-free survival (RRFS) | 5 years
  RRFS is defined as the time period between registration and first regional event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
brain metastasis free survival (in the subgroup of TNBC and HER2+) | 5 years
  brain metastasis free survival is defined as the time period between registration and first brain metastasis event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
compliance | 5 years
  compliance is defined as the adherence to protocol and will be analyzed after the end of the therapy by referring to data from CRF.
safety | 5 years
  safety is defined by the AE that occur and will be analyzed after the end of the therapy by referring to data from CRF (including time to resolve neuropathy to grade 1)
side effects of taxane | 5 years
  Side effects of taxane are measured before, during and after chemotherapy by FACT-taxane questionnaires. the questionnaires will be analyzed after the end of the therapy.
treatment effects by intrinsic subtypes | 5 years
  the treatment effect will be analyzed after the end of the therapy by referring to data from CRF and later by using the data from patient registry to compare the outcome in the different subtypes. The intrinsic subtypes are: 0-3, 4-9 or 10+ involved nodes as well as Ki-67.
Ovarian substudy | Baseline, 6 months, 12 months, 18 months, 24 months 30 months
  To assess ovarian function measured by amenorrhea rate in correlation with changes in E2, FSH, LH , Anti-Müller Hormone, ultrasound-follicle count in patients aged <45 years.
Pharmacogenetic substudy | Baseline
  To correlate Single Nucleotide Polymorphisms (SNPs) of genes with the associated toxicity and histologically assessed treatment effect.
biology of lymph node metastases | baseline
  The correlation of lymph node metastases with biological markers is investigated

OTHER OUTCOMES:
prognostic/predictive factors | 5 years
  the treatment effect will be analyzed after the end of the therapy by referring to data from CRF and later by using the data from patient registry to correlate the outcome with biological markers.

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, Prof., Study Chair — GBG Forschungs GmbH
Locations (1):
- Klinikum Frankfurt Höchst, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Denkert C, Seither F, Schneeweiss A, Link T, Blohmer JU, Just M, Wimberger P, Forberger A, Tesch H, Jackisch C, Schmatloch S, Reinisch M, Solomayer EF, Schmitt WD, Hanusch C, Fasching PA, Lubbe K, Solbach C, Huober J, Rhiem K, Marme F, Reimer T, Schmidt M, Sinn BV, Janni W, Stickeler E, Michel L, Stotzer O, Hahnen E, Furlanetto J, Seiler S, Nekljudova V, Untch M, Loibl S. Clinical and molecular characteristics of HER2-low-positive breast cancer: pooled analysis of individual patient data from four prospective, neoadjuvant clinical trials. Lancet Oncol. 2021 Aug;22(8):1151-1161. doi: 10.1016/S1470-2045(21)00301-6. Epub 2021 Jul 9. PMID 34252375